CLINICAL TRIAL: NCT05018624
Title: Alcohol Brief Intervention Integrated With Mobile Chat-based Support for Risky Drinkers in Emergency Departments: a Pragmatic Randomised Controlled Trial
Brief Title: Alcohol Brief Intervention Integrated With Mobile Chat-based Support for Risky Drinkers in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chat-based ABI (AED)
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Misuse
Keywords: Chat-based IM; Alcohol brief intervention; AED; AUDIT
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Alcohol brief intervention, leaflets, regular personalized messages on ABI through IM Apps, real-time chat-based support through IM Apps
  Interventions: Behavioral: Alcohol brief intervention; Behavioral: 12-page health warning leaflet; Behavioral: Regular messages through Instant Messaging (IM); Behavioral: Real-time chat-based support through IM Apps; Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong
- control group (Active Comparator): Alcohol brief intervention, leaflets, regular messages on general health through SMS
  Interventions: Behavioral: Alcohol brief intervention; Behavioral: 12-page health warning leaflet; Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong

INTERVENTIONS:
Behavioral: Alcohol brief intervention — At baseline, subjects will receive face-to-face or online alcohol brief intervention developed based on the guideline by the World Health Organisation in 5-10 minutes
Behavioral: 12-page health warning leaflet — Nurses will provide information about the consequences of drinking using a 12-page health warning booklet. Benefits of reducing and quit drinking will be emphasized by focusing on improving their perception towards the impacts on health, social problems, risky behaviors, academic performance and financial issues.
Behavioral: Regular messages through Instant Messaging (IM) — A total of 26 e-messages will be scheduled: once daily for the first week, 3 time/week for subsequent 4 weeks and 1 time/week for the remaining 7 weeks. The frequency will be adjusted according to IM Apps conversation and subject's requests.
  Arms: Intervention group
Behavioral: Real-time chat-based support through IM Apps — The chat-based IM support is the extension of baseline ABI and regular e-messages, which aims to provide real-time behavioral and psychosocial support to reduce or quit drinking. It will be personalized according to the subjects' characteristics (gender, drinking pattern and alcoholic drinks preferences), intention to drink and specific questions regarding drinking. Through real-time chatting (text and/or voice), drinkers can acquire information on consequences of drinking and gain social support immediately to reduce intention to drink and alcohol consumption.
  Arms: Intervention group
Behavioral: AUDIT score interpretation sheet adapted from the Department of Health of Hong Kong — a diagram explaining drinking behaviour and potential health risks, definitions of "alcohol unit" and "binge drinking", and advise on limiting daily drinking to 2 alcohol units for men and 1 unit for women

SUMMARY:
This study aims to assess the effectiveness of chat-based intervention on reducing risky alcohol consumption to inform clinical practice for providing ABI to risky drinkers attending AED in Hong Kong.

DETAILED DESCRIPTION:
Alcohol use is a major risk factor for non-communicable diseases and 6th leading cause of death and disability-adjusted life years. The prevalence of alcohol consumption has increased since 2008 after introduction of zero tax on alcohol with strength <30% (e.g., wine and beer) and due to promoting the city as Asia's wine hub. ABI reduced alcohol intake by about 20g/week at 12-month follow-up in primary healthcare populations. Given the relatively low prevalence of risky alcohol drinkers in Hong Kong, testing ABI in clinics may face difficulties in recruitment. Alcohol use is associated with problems such as injury and violence requiring accident and emergency department (AED) services, thus AEDs in Hong Kong are more feasible places to recruit subjects for delivering ABI.

Primary hypothesis: The Intervention group has significantly larger reduction of weekly alcohol consumption compared with the Control group at 12-month follow-up

Secondary hypotheses: Compared with the Control group, the Intervention group has lower AUDIT scores, fewer episodes of heavy/binge drinking, lower re-attendence at AED and reduced alcohol-related harms at 6-month and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HK resident able to read/communicate in Cantonese/Putonghua. This may exclude potential subjects from other countries with higher alcohol consumption than local Chinese, but quality of the chat-based intervention is important for the research hypothesis, and it will not be feasible to recruit other language speakers (e.g., English) in the present study.
* Aged ≥18 with proficiency in using IM Apps (e.g., WhatsApp, WeChat). Those aged <18 are excluded as other studies suggest they have different patterns of alcohol drinking and reduction from adult drinkers.

Exclusion Criteria:

* Those unable to understand or receive face-to-face ABI due to severe traumatic injury, unconscious, or drunk patients unable to follow commands
* Anticipated to be admitted to in-patient department for >1 week, which will interfere with the chat-based intervention
* Having psychiatric/psychological diseases or receiving regular psychotropic medication
* Participating in other alcohol reduction or abstinence programmes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Amount of alcohol consumption per week (gram/week) at 12-month follow-up | 12-month after baseline
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 12-month after baseline.
Compare the primary outcome using intention-to-treat (ITT), per-protocol (PP) and as-treated (AP) analysis with Compliance Average Causal Effect (CACE) analysis | 6-month after baseline
  To estimate large, moderate and null (same as the control) treatment effects and check whether ITT, AP and PP analysis estimates are biased compared with CACE estimates (alcohol consumption per week at 6-month follow-up)

SECONDARY OUTCOMES:
Amount of alcohol consumption per week (gram/week) at 3- and 6-month follow-ups | 3 and 6 months after baseline
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 3- and 6-month after baseline.
AUDIT scores at 3-, 6- and 12-month follow-ups | 3, 6 and 12 months after baseline
  Assessed by Alcohol Use Disorders Identification Test (ranged 0-40 with higher score indicating problematic alcohol use) and compare the AUDIT between intervention and control group at 3-, 6- adn 12-month after baseline.
Number of standard drinks (10g of alcohol) per week at 3-, 6-, and 12-month follow-ups | 3, 6 and 12 months after baseline
  Assessed by either increase or decrease in standard drinks number and compared between intervention and control group at 3-, 6-, and 12-month
Episode of binge drinking in the past 30-day at 3-, 6- and 12-month follow-ups | 3, 6, and 12 months after baseline
  Defined by 5 standard drink [male] or 4 standard drink [female] in one occasion for binge drinking and compared between intervention and control group at 3-, 6-, and 12-month
Episode of heavy drinking in the past 30-day at 3-, 6- and 12-month follow-ups | 3, 6, and 12 months after baseline
  Defined by 15 standard drink [male] or 8 standard drink[female] in a week for heavy drinking and compared between intervention and control group at 3-, 6-, and 12-month
Planned drinking measured in the coming 30-day at 3-, 6- and 12-month follow-ups | 3, 6, and 12 months after baseline
  Compare the number of planned drinking (yes or no) between intervention group and control group at 3-, 6- and 12-month follow-ups
Re-attendance of AED at 3-, 6- and 12-month follow-ups | 3, 6, and 12 months after baseline
  Ask for attendance of AED (yes/no) in the past 3 months at 3-, 6- and 12-month follow-ups
Health status of participants at 12-month | 12 months after baseline
  Measured by EQ-5D-5L. Comprises five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION), each dimension has five response levels:no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The participant is asked to indicate his/her health state by checking the box next to the most appropriate response level. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. Extreme problem is coded as 5, severe problem is coded as 4, moderate is coded as 3, slight problem is coded as 2 and no problem is coded as 1.
Current health of participants at 12-month | 12 months after baseline
  Measured by EQ VAS. Participant is asked to rate his/her health on a vertical visual analogue scale. The scale is numbered from 0-100.100 means the best health, 0 is the worst. Participant will put a "cross" on the scale to indicate his/her current health.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong